CLINICAL TRIAL: NCT03580551
Title: Older Veterans EmpoweRed To Use Regular Exercise (OVERTURE) II
Acronym: OVERTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Karlene K Ball, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-300001897
Record Dates: First submitted 2018-06-12; First posted 2018-07-09 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Quality of Life; Aging
Keywords: Veterans; Sedentary; Chronic illness
MeSH Terms: conditions — Sedentary Behavior; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Ten participants from each racial group (Black/White) will be assigned to the Intervention, which will receive the home-based DVD Chair Exercise Program. This is the group that will receive the chair exercise intervention upon enrollment.
  Interventions: Behavioral: Intervention Group
- Waitlist Control Group (Active Comparator): Ten participants from each racial group (Black/White) will be assigned to the Waitlist Control Group, which will receive the home-based DVD Chair Exercise Program at the end of 8 weeks.
  Interventions: Behavioral: Waitlist Control Group

INTERVENTIONS:
Behavioral: Intervention Group — Intervention group participants will receive the home-based DVD chair exercise program, which will include a DVD player, "Sit and Be Fit" DVD, schedule of exercise sessions, hand weights, exercise balls, resistance bands, exercise log, and satisfaction survey. Participants will be instructed to complete an assigned "Sit and Be Fit" exercise session once a day (sessions last approximately 30 minutes), five days a week (Monday-Friday) for 8 weeks. During the first 6 weeks, the intervention group will not have contact with the study team, unless to trouble-shoot the DVD or answer questions about exercise sessions. At the end of week 6, the intervention group will be contacted to schedule a post-assessment for the end of week 8, which will include repeating all health measures, except for health status.
  Arms: Intervention Group
Behavioral: Waitlist Control Group — At week 8, waitlist control group will receive the home-based DVD chair exercise program, which will include a DVD player, "Sit and Be Fit" DVD, schedule of exercise sessions, hand weights, exercise balls, resistance bands, exercise log, and satisfaction survey. The waitlist control group will complete a post-assessment at the end of week 8, which will include all health status measures, except health status. Waitlist control group will be instructed to complete an assigned "Sit and Be Fit" exercise session once a day (sessions last approximately 30 minutes), five days a week (Monday-Friday) for 8 weeks. Waitlist control group will not have contact with the study team, unless to trouble-shoot the DVD or answer questions about exercise sessions. At the end 14 weeks, waitlist control group will be contacted to schedule a final meeting, and to collect the adherence logs and satisfaction survey. At 16 weeks, the waitlist control group will not receive an additional post-assessment.
  Arms: Waitlist Control Group

SUMMARY:
The purpose of this study is to investigate the practicality of a short-term (8-weeks), home-based digital versatile disc (DVD) chair exercise program among 40 sedentary older Black/African American and White/Caucasian veterans with three or more chronic health conditions, such as type 2 diabetes, hypertension, and osteoarthritis.

DETAILED DESCRIPTION:
This study will determine the feasibility of a home-based DVD chair exercise program, "Sit and Be Fit." Participants will be asked to complete a chair-exercise program Monday through Friday. Each chair exercise session lasts approximately 30 minutes. Participants will receive a new DVD player, the exercise DVD, and the necessary exercise equipment to complete each session. The equipment includes a set of 1 pound hand weights, a 10" exercise ball, a small handball, a resistance band, an exercise log, and a satisfaction survey. Upon initial enrollment, both groups will receive a baseline health assessment that will include health-related quality of life, subjective well-being, body mass index (BMI), comorbidity, blood pressure, lower body extremity fitness, physical activity, and hand grip strength. Excluding health status, all other measures will be completed at post-assessment (the end of week 8 for Group A and Group B). The intervention group (Group A) will receive the equipment after completing eligibility screening, an informed consent, and health assessments. The waitlist control group (Group B) will receive the equipment at week 9 after the post-assessment. Group B will complete the program through week 16. The waitlist control group(Group B) will not receive an additional post assessment at the end of week 16.

ELIGIBILITY:
Inclusion Criteria:

* Be a veteran, which will be verified through documentation, such as discharge papers, military identification card, or military photographs
* Identify as Black/African American or White/Caucasian; demonstrate proof of age 65+; self-report of three or more chronic health conditions
* Pass a cognitive screening related to thinking/reasoning/decision making; report less than 30 minutes of daily physical activity
* Systolic blood pressure lower than 180
* Diastolic blood pressure lower than 100
* Resting heart rate 90 or lower
* Three or more chronic health conditions
* Permission from primary care physician (PCP)
* Own a sturdy stand-alone chair without arms
* Own an operable television
* Willing to be randomized to the intervention or the waitlist control group

Exclusion Criteria:

* Non-veteran
* Non-Black or African American/White or Caucasian
* Younger than 65 years of age
* Systolic blood pressure 180 or higher
* Diastolic blood pressure is 100 or higher
* Resting heart rate higher than 90
* Less than three chronic health conditions
* Failure to pass a cognitive screening
* Report more than 30 minutes of daily physical activity
* No approval from PCP
* No sturdy stand-alone chair without arms
* No operable television
* Unwilling to be assigned to the intervention or the waitlist control group

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Number of fitness sessions completed based on participants' activity logs - Adherence to the home-based DVD chair exercise program | At the end of 8 weeks.
  Adherence (number of fitness sessions completed based on participants' activity logs). Participants' activity logs will be used to assess subjective completion of fitness sessions.
Number of participants lost to attrition | At the end of 8 weeks.
  The number of participants lost to attrition (dropped out). This will be measured by the number of participants that have completed the entire 8 week program. Before and after each session, participants will be instructed to record the date and time the session was started and completed.
Participants' program satisfaction | At the end of 8 weeks.
  Satisfaction ratings will be assessed based on participants' satisfaction logs.
Participants' rating of the program | Week 10
  Intervention group participants' ratings of the intervention based on open-ended questions asked during the focus group session.

SECONDARY OUTCOMES:
To evaluate the Quality of Life (QOL) of participants | Baseline and post-assessment at week 8.
  The 36-Item Short Form Survey (SF-36) will be used to assess QOL outcomes. A 0 score indicates the lowest level of QOL measured by the scale and a 100 indicates the highest level of QOL measured by the scale.
Subjective Well-being (SWB) | Baseline and post-assessment at week 8.
  How an individual rates general feelings of happiness (well-being). SWB will be measured using a modified SWB scale. The scale consists of 4 items that assess overall happiness. Respondents were asked two questions about their happiness as well as two questions comparing their happiness to the happiness of others on a scale from 1 to 7, with 7 reflecting a high degree of perceived happiness. Composite scores on the scale range from 4 to 28.
Physical Activity | Baseline and post-assessment at week 8.
  The Physical Activity Scale for the Elderly (PASE) will be used to assess level of physical activity. Score ranges from 0 to 360. A high score indicates a high level of physical activity.
Blood pressure | Baseline and post-assessment at week 8
  Blood pressure (systolic and diastolic) will be assessed using a standard blood pressure cuff.
Heart Rate (Pulse) | Baseline and post-assessment at week 8
  Pulse rate will be assessed using a standard blood pressure cuff.
Body Mass Index (BMI) | Baseline and post-assessment at week 8.
  BMI will be assessed using a standard weight scale and a folding yardstick.
Hand Grip Strength | Baseline and post-assessment at week 8.
  Hand grip strength will be assessed using a Baseline Hydraulic Hand Dynamometer.
Short Physical Performance Battery (SPPB) | Baseline and post-assessment at week 8.
  The SPPB will assess lower body function with a balance test, gait (walk) test, and chair stands.
Comorbidity | Baseline
  Comorbidity will be assessed using the Charlson Comorbidity Index. Comorbidity is the presence of additional chronic health conditions that can impact life expectancy. Individual chronic conditions will be assigned a score based on severity and averaged. Based on the chronic condition, assigned scores can be 1, 2, 3, or 6.

CONTACTS AND LOCATIONS:
Overall Officials: Karlene K Ball, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] McCaskill GM, Clay OJ, Motl RW, Ball KK. Older Veterans EmpoweRed To Use Regular Exercise (OVERTURE) II: Design and methods of a randomized controlled trial among older veterans with chronic health conditions. Contemp Clin Trials Commun. 2019 Jun 28;15:100395. doi: 10.1016/j.conctc.2019.100395. eCollection 2019 Sep. No abstract available. PMID 31338477